CLINICAL TRIAL: NCT05902247
Title: Phase I Dose Escalation Study to Evaluate Tolerability and Safety of 225Ac-PSMA I&T in Patients With Metastatic Prostate Cancer
Brief Title: Actium-225-Prostate Specific Membrane Antigen Imaging & Therapy
Acronym: 225AcPSMAI&T
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Tessa Brabander, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL73234.078.20
Record Dates: First submitted 2023-05-24; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: 225Ac-PSMA; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: A clinical prospective, single-center, single-arm, phase I dose escalation therapy study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 225Ac-PSMA I&T (Experimental): 225Ac-PSMA I&T
  Interventions: Radiation: Radionuclide Therapy

INTERVENTIONS:
Radiation: Radionuclide Therapy — To evaluate the tolerability and safety of 225Ac-PSMA I&T in patients with metastatic prostate cancer
  Other Names: 225Ac-PSMA I&T

SUMMARY:
225Ac-PSMA I&T is a radiopharmaceutical for therapy of prostate cancer. PSMA is overexpressed on prostate cancer cells. Actium-225 is an alpha emitting radionuclide. When PSMA I&T is labelled with Actium-225, it can be applied as therapy for prostate cancer.

DETAILED DESCRIPTION:
Rationale:

225Ac-PSMA I&T is a radiopharmaceutical for therapy of prostate cancer. PSMA is overexpressed on prostate cancer cells. Actium-225 is an alpha emitting radionuclide. When PSMA I&T is labelled with Actium-225, it can be applied as therapy for prostate cancer.

Objective:

To evaluate the tolerability and safety of 225Ac-PSMA I&T in patients with metastatic prostate cancer and recommend a dose for further phase 2 studies.

Study design:

A clinical prospective, single-center, single-arm, phase I dose escalation therapy study.

Study population:

Up to 30 patients with advanced metastatic castration-resistant prostate cancer (mCRPC).

Intervention:

Patients with advanced mCRPC will receive therapy with 225Ac-PSMA I&T. The first dose-level will not exceed 8 megabecquerel (MBq), as this is reported in the literature as a save activity for treatment. A Positron Emission Tomography - Magnetic Resonance Imaging (PET-MRI) with Gallium-68-PSMA I&T (68Ga) will be performed to calculate the precise dose-level needed and as a verification the precise dose-level will be compared with the dose-level of 8 MBq. In the first week after therapy, the PET-MRI will be repeated to observe any effects of the alpha radiation on the metastases and observe the potential changes in 68Ga-PSMA I&T uptake. Eight weeks after the first cycle, patients will receive the second cycle of 225Ac-PSMA I&T. If no Dose Limiting Toxicity (DLT) occurs, the dose can be increased for the next DL. If a DLT occurs, the cohort will be expanded to 6 patients. After establishing the recommended dose, an expansion cohort will be opened with a total of 12 patients.

Main study endpoints:

To investigate the safety, tolerability and biochemical effects of 225Ac-PSMA I&T injected in patients with metastatic prostate cancer.

Primary objective:

- To assess the safety and tolerability of 225Ac-PSMA I&T administered intravenously

Secondary objectives:

* To predict and calculate the absorbed-dose in critical organs (e.g. salivary glands, kidneys, bone marrow) by 68Ga-PSMA I&T PET-MRI
* To evaluate the effects of the radionuclide therapy on metastases in the days after therapy using 68Ga-PSMA I&T PET-MRI
* To evaluate the biochemical effects of 225Ac-PSMA I&T therapy in patients with metastatic prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Histopathological proven metastatic castration resistant prostate cancer. Castrationresistant disease is defined as a serum testosterone level of 50 nanogram per deciliter or lower (≤1.7 nanomol per liter) after bilateral orchiectomy or during maintenance treatment consisting of androgen-ablation therapy with a luteinizing hormone-releasing hormone agonist.
* Evidence of progressive disease, defined as 1 or more Prostate Cancer Work Grouping 3 (PCWG3) criteria: - PSA level ≥ 1 ng/mL that has increased on at least 2 successive occasions at least 1 week apart
* Progression as defined by RECIST 1.1 with PCGW3 modifications
* Progression after at least one line of chemotherapy and/or one line of nonsteroidal antiandrogen (NSAA).
* No active anti-tumor therapy, except for androgen deprivation therapy in combination with at least one androgen receptor-targeted agent
* Willing and able to undergo 2 cycles of 225Ac-PSMA I&T therapy and 3 PET-MRI scans in 16 weeks and comply with protocol
* Signed and dated written informed consent by the patient (or legal representative) prior to any study-specific procedures.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance-status score 0-2.
* Use of highly effective methods of contraception (female partners of male participants)
* During the trial and 6 months after completion of the study or willing to practice sexual abstinence.

Exclusion Criteria:

* Concurrent severe illness or clinically relevant trauma within 2 weeks before the administration of the investigational product that might preclude study completion or interfere with study results
* Serum hemoglobin ≤ 6.2 mmol/L, total white blood cell (WBC) count ≤ 3.5·109/L, absolute neutrophil count ≤ 1.5·109/L, platelet count ≤ 100·109/L, serum creatinine concentration ≥ 150 umol/L (≥ 1.7 mg/dL), serum albumin <30 g/L, bilirubin ≥ 1.5 x upper limit normal (ULN), aspartate transaminase (ASAT) ≥ 3 x ULN and alanine aminotransferase (ALAT) ≥ 3 x ULN (or bilirubin ≥ 3 x ULN, ASAT ≥ 5 x ULN and ALAT ≥ 5 x ULN in the case of pre-existing liver metastases at baseline)
* Concurrent bladder outflow obstruction or unmanageable urinary incontinence
* Known or expected hypersensitivity to Gallium-68, Actinium-225, PSMA I&T, or any excipient present in 225Ac/68Ga-PSMA I&T
* Prior administration of a radiopharmaceutical within a period corresponding to 8 halflives of the radionuclide used on such radiopharmaceutical
* Prior treatment with any radionuclide therapy
* History of somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study
* Central nervous system (CNS) metastases, leptomeningeal disease, or spinal cord compression
* Radiation therapy within 4 weeks of first dose (or local or focal radiotherapy within 2 weeks of first dose)
* Male subjects unwilling to abstain from donating sperm during treatment and for an additional 6 months after the last dose

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 30 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events and Serious Adverse Events as assessed by CTCAE v5.0 | 4 years
  Safety and tolerability assessment
Absolute values and changes from baseline in laboratory parameters (hematology, blood chemistry and urinalysis), including assessment of shifts from baseline to abnormal values on treatment | 4 years
  Safety and tolerability assessment
Absolute values and changes from baseline in vital signs & ECG parameters | 4 years
  Safety and tolerability assessment

SECONDARY OUTCOMES:
To predict and calculate the absorbed-dose in critical organs (e.g. salivary glands, kidneys, bone marrow) by 68Ga-PSMA I&T PET-MRI | 4 years
  Dosimetry
Changes in SUVmax of the target lesions on PET-MRI and morphological changes evaluated on MRI | 4 years
  Direct effect of 225Ac-PSMA I&T
Objective response rate (ORR) as measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria v.1.1. | 4 years
  Preliminary efficacy
Percent changes from baseline in tumor size where tumor size is defined as the sum of all target lesions as measured by RECIST criteria v.1.1. | 4 years
  Preliminary efficacy
Prostate Specific Antigen(PSA) response rate assessed from treatment visit 1 defined as a decrease in PSA of ≥ 50% from baseline. | 4 years
  Preliminary efficacy
Percent change from baseline in PSA as a continuous endpoint by visit and maximum reduction during the study | 4 years
  Preliminary efficacy
Percent change from baseline values of pain questionnaire at every treatment visit | 4 years
  Preliminary efficacy
Overall Survival (OS) defined as the time from the date of first dose of 225Ac-PSMA I&T treatment to the date of death due to any cause. | 4 years
  Preliminary efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ling SW, van der Veldt AAM, Konijnenberg M, Segbers M, Hooijman E, Bruchertseifer F, Morgenstern A, de Blois E, Brabander T. Evaluation of the tolerability and safety of [225Ac]Ac-PSMA-I&T in patients with metastatic prostate cancer: a phase I dose escalation study. BMC Cancer. 2024 Jan 29;24(1):146. doi: 10.1186/s12885-024-11900-y. PMID 38287346